CLINICAL TRIAL: NCT05911451
Title: Optimizing Access Surgery In Senior Hemodialysis Patients: a Multicenter Randomized Controlled Trial of Fistulas, Grafts, and Catheters
Brief Title: Optimizing Access Surgery In Senior Hemodialysis Patients
Acronym: OASIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL70385.068.19; NL7933 (Other: Netherlands Trial Registry)
Record Dates: First submitted 2023-05-26; First posted 2023-06-22 (Actual); Last update posted 2025-05-19 (Actual); Status verified 2025-05

CONDITIONS: Vascular Access Complication; Hemodialysis Access Failure; Dialysis Access Malfunction; Arteriovenous Fistula; Arteriovenous Graft; Central Venous Catheter Related Bloodstream Infection
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Central Venous Catheters

STUDY DESIGN:
Intervention Model Description: Parallel group, multicenter randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arteriovenous fistula (Active Comparator): Patients allocated to usual care will be treated according to current guidelines on vascular access creation. These guidelines recommend placing autologous arteriovenous fistulas at the most distal site with adequate blood vessels, preferably in the non-dominant arm. Patients who have already been on hemodialysis treatment using a central venous catheter must be operated within 6 months of dialysis initiation. Because the study aims to compare the different surgical strategies for vascular access creation in a real-life situation, the study will not interfere with clinical practice at the study sites.
  Interventions: Procedure: Arteriovenous fistula creation
- Arteriovenous graft (Experimental): Patients who are allocated to the arteriovenous graft strategy will have a commercially available prosthetic tube graft implanted for hemodialysis access. Patients who have already been on hemodialysis treatment using a central venous catheter must be operated within 6 months of dialysis initiation. Because the study aims to compare the different surgical strategies for vascular access creation in a real-life situation, the study will not interfere with clinical practice at the study sites.
  Interventions: Procedure: Arteriovenous graft placement
- Central venous catheter (Experimental): Patients who are allocated to the central venous catheter strategy will have a dialysis catheter inserted. Because the study aims to compare the different surgical strategies for vascular access creation in a real-life situation, the study will not interfere with clinical practice at the study sites.
  Interventions: Procedure: Central venous catheter placement

INTERVENTIONS:
Procedure: Arteriovenous fistula creation — It is recommended to create the arteriovenous fistula 3 to 6 months before the expected start of hemodialysis treatment using locoregional anesthesia. It is recommended to use minimal venous and arterial diameters of 2mm for radiocephalic fistulas and 3mm for brachiocephalic and brachiobasilic fistulas. It is recommended to avoid creating an arteriovenous fistula at the same side as a pacemaker, central venous catheter, or arterial stenosis. It is recommended to use the following order of preference for arteriovenous fistula creation: radiocephalic fistula as first choice, brachiocephalic fistula as second choice, and brachiobasilic fistula as third choice.
  Arms: Arteriovenous fistula
Procedure: Arteriovenous graft placement — It is recommended to implant the arteriovenous graft 2 weeks before the expected start of hemodialysis treatment under antibiotic prophylaxis. Implantation of an early-cannulation graft is recommended for patients who require more urgent start of hemodialysis to avoid the use of a temporary central venous catheter. It is recommended to use minimal arterial and venous diameters of 3mm and 4mm, respectively. It is recommended to avoid placing an arteriovenous graft at the same side as a pacemaker, central venous catheter, or arterial stenosis.
  Arms: Arteriovenous graft
Procedure: Central venous catheter placement — It is recommended to place a tunneled central venous catheter just before the start of hemodialysis treatment under local anesthesia, with conscious sedation if preferred by the patient. The catheter should preferably be placed in the right internal jugular vein with ultrasound-guided puncture and fluoroscopy control under sterile conditions. According to usual practice at the trial center, catheters may be implanted by surgeons, interventional radiologists, or nephrologists.
  Arms: Central venous catheter

SUMMARY:
The number of elderly hemodialysis patients is growing. Vascular access complications are a major determinant of the quality of life and health care costs for these vulnerable patients. The three different types of vascular access, i.e. autologous arteriovenous fistulas, arteriovenous grafts, and central venous catheters, have never been compared in randomized controlled trials. This project will deliver the much-needed evidence to determine the optimal strategy for vascular access creation in elderly hemodialysis patients in order to deliver better health care at lower costs.

DETAILED DESCRIPTION:
Objective: To compare surgical strategies for vascular access creation in elderly hemodialysis patients.

Hypothesis: Arteriovenous grafts and central venous catheters lead to fewer interventions, more quality of life, and lower health care costs than autologous arteriovenous fistulas.

Study design: Parallel group, multicenter randomized controlled trial.

Study population: Patients >65 years with a life expectancy <2 years who are expected to start hemodialysis treatment within 6 months or who have started hemodialysis treatment with a catheter in the past 6 months.

Study groups:

1. Autologous arteriovenous fistula creation
2. Arteriovenous graft implantation
3. Central venous catheter placement

Sample size calculation: 3x65 patients for superiority with multiplicity correction based on a clinically relevant difference of 0.80 interventions/year. Due to slow enrollment, follow-up time per participant was much longer than anticipated at trial initiation. After enrollment of 166 participants, calculations based on actual event and mortality rates showed that the trial had sufficient statistical power to detect a relative difference in event rate of 0.67, corresponding to an absolute difference below the minimal clinically relevant difference of 0.80 access-related interventions per year. Therefore, enrollment was closed at 166 participants.

Data analysis: Poisson regression analysis with time as off-set variable.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 65 years or older
2. End-stage renal disease with unlikely recovery of kidney function according to the attending nephrologist
3. Hemodialysis is the intended long-term modality of treatment for end-stage renal disease
4. Fit for vascular access surgery as determined by the local multidisciplinary vascular access team 5a. Expected to start hemodialysis treatment within 6 months at the time of treatment assignment; or 5b. Treated with hemodialysis for 6 months or less at the time of treatment assignment using a tunneled or non-tunneled central venous catheter for vascular access

6. Planning to remain in one of participating dialysis centers for at least 1 year 7. Suitable vascular anatomy for all types of vascular access based on duplex ultrasound of the arms, defined as:

* at least one suitable configuration for an arteriovenous fistula using minimal arterial and venous diameters of 2mm for radiocephalic fistulas and 3mm for brachiocephalic and brachiobasilic fistulas;
* at least one suitable configuration for an arteriovenous graft using minimal arterial and venous diameters of 3mm and 4mm, respectively; and
* at least one open internal jugular vein for a central venous catheter.

Exclusion Criteria:

1. Patent arteriovenous fistula or graft already in place
2. Prior unsuccessful arteriovenous fistula or graft vascular access surgery
3. Kidney transplantation planned within 6 months
4. Metastatic malignancies or other condition associated with a life expectancy of <6 months, in the opinion of the attending nephrologist
5. Unable to provide informed consent
6. Dusseux risk score <5, indicating an usually long life expectancy for elderly patients starting hemodialysis treatment (the Dusseux risk score was adapted for patients between 65 and 70 years by assigning -3 points to this age category)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 166 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Access-related intervention rate | Variable follow-up time of at least 1 year
  The number of access-related interventions required for each person-year of hemodialysis treatment. This outcome measure includes all percutaneous access interventions (including central venous catheter placement, removal and guidewire exchange, angioplasty, stent placement, and percutaneous thrombectomy) and surgical access procedures (including initial access creation, subsequent access placements if the first access failed, and surgical revisions to promote maturation or maintain long-term patency, including open thrombectomy) from randomization and treatment assignment until the end of the study period or death.

SECONDARY OUTCOMES:
Patient-reported outcome measures (1) | Every 3 months in the first year after enrollment and in the first year after dialysis start
  Short Form 12 Dialysis Symptom Index (SF-12 / DSI)
Patient-reported outcome measures (2) | Every 3 months in the first year after enrollment and in the first year after dialysis start
  Short Form Vascular Access Questionnaire (SF-VAQ)
Patient-reported outcome measures (3) | Every 3 months in the first year after enrollment and in the first year after dialysis start
  EuroQol - 5 dimensions - 5 levels (EQ-5D-5L)
Health care costs | Every 3 months in the first year after enrollment and in the first year after dialysis start
  Medical Consumption Questionnaire
Access-related complications | Variable follow-up time of at least 1 year
  Access-related complications requiring pharmacological treatment (Clavien-Dindo grade 2)
Days in hospital | Variable follow-up time of at least 1 year
  The number of days admitted to hospital or visiting out-patient clinics for any reason per person-year (including hemodialysis sessions).
Mortality | Variable follow-up time of at least 1 year
  All-cause mortality
Primary patency | Variable follow-up time of at least 1 year
  Outcome measure registered for exploratory analysis
Assisted primary patency | Variable follow-up time of at least 1 year
  Outcome measure registered for exploratory analysis
Secondary patency | Variable follow-up time of at least 1 year
  Outcome measure registered for exploratory analysis
Primary functional patency | Variable follow-up time of at least 1 year
  Outcome measure registered for exploratory analysis
Time until mature vascular access | Variable follow-up time of at least 1 year
  Outcome measure registered for exploratory analysis
Time until functional vascular access | Variable follow-up time of at least 1 year
  Outcome measure registered for exploratory analysis
The number of hemodialysis sessions with cannulation difficulties | Variable follow-up time of at least 1 year
  Outcome measure registered for exploratory analysis

CONTACTS AND LOCATIONS:
Overall Officials: Maarten G Snoeijs, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (20):
- Netherlands (20):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - OLVG, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Spaarne Gasthuis, Haarlem
  - Zuyderland Medisch Centrum, Heerlen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Haaglanden Medisch Centrum, The Hague
  - Elisabeth Tweesteden Ziekenhuis, Tilburg
  - Maxima Medisch Centrum, Veldhoven
  - Viecuri Medisch Centrum, Venlo
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
The following end products I will make available for further research and verification:
  * Data documentation
  * Documentation of the research process, including documentation of all participants
  * Audiovisual material / images
  * Several versions of processed data
  * Raw data
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The embargo period will be as long as required for publication of the research findings.
Access Criteria: Interested parties can submit a request for a data set.